CLINICAL TRIAL: NCT02203630
Title: A Randomized Controlled Pilot Trial of Phenylephrine Versus Norepinephrine for Septic Shock in Critically Ill Patients
Brief Title: Phenylephrine Versus Norepinephrine for Septic Shock in Critically Ill Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment; Lack of support and equipoise
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 140141; UL1RR024975-01 (NIH); UL1TR000445-06 (NIH)
Record Dates: First submitted 2014-07-22; First posted 2014-07-30 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-05

CONDITIONS: Septic Shock; Sepsis; Shock; Tachycardia; Arrhythmia
Keywords: Septic shock; Vasopressor Agents; Phenylephrine; Norepinephrine; Tachycardia; Heart Rate; Arrhythmia; Catecholamine
MeSH Terms: conditions — Shock, Septic; Sepsis; Shock; Tachycardia; Arrhythmias, Cardiac | interventions — Phenylephrine; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenylephrine (Active Comparator): Phenylephrine will be administered as the primary vasopressor for the treatment of septic shock
  Interventions: Drug: Phenylephrine
- Norepinephrine (Active Comparator): Norepinephrine will be administered as the primary vasopressor for the treatment of septic shock
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Phenylephrine — Phenylephrine, in intravenous formulation, will be administered as the primary vasopressor for the treatment of septic shock
  Other Names: Neosynephrine
  Arms: Phenylephrine
Drug: Norepinephrine — Norepinephrine, in intravenous formulation, will be administered as the primary vasopressor for the treatment of septic shock
  Other Names: Levophed
  Arms: Norepinephrine

SUMMARY:
Septic shock is a condition that is marked by severe infection causing hypotension requiring vasopressors to maintain adequate perfusion to vital organs. The Surviving Sepsis campaign, an international organization formed for the purpose of guiding the management of sepsis and septic shock, currently recommends norepinephrine as the first-choice vasopressor for septic shock. Phenylephrine, a vasopressor FDA-approved for use in septic shock, is recommended as an alternative vasopressor when septic shock is complicated by tachyarrhythmia to mitigate cardiac complications. This recommendation is based solely on experience with no scientific evidence to support this recommendation.

The investigators will conduct an open-label randomized controlled trial (RCT) directly comparing phenylephrine and norepinephrine, two FDA-approved vasopressors that are both used in clinical practice for the management of septic shock. The investigators will perform this study with a population of patients that have septic shock to complete the following aims:

Aim 1: Determine the incidence of tachyarrhythmias.

Aim 2: Determine which vasopressor, phenylephrine or norepinephrine, is associated with a lower heart rate.

Aim 3: Determine which vasopressor, phenylephrine or norepinephrine, is associated with a higher incidence of new tachyarrhythmias.

Aim 4: Determine which vasopressor, phenylephrine or norepinephrine, is associated with less time in tachyarrhythmia.

Aim 5: Determine which vasopressor, phenylephrine or norepinephrine, is associated with fewer complications, including cardiac complications.

The investigators hypothesize that in this setting, phenylephrine will improve the management of septic shock when used as a "first choice" vasopressor by:

1. Decreasing the mean heart rate
2. Decreasing the incidence of new tachyarrhythmias
3. Decreasing the amount of time spent in tachyarrhythmia for patients who develop new onset and recurrent tachyarrhythmias
4. Decreasing the number of cardiac complications

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or greater
* Intention to treat with vasopressor for diagnosis of septic shock
* Exclusion criteria not met

Exclusion Criteria:

* Emergent indication for surgery
* Patient possesses a terminal condition for which patient or medical decision maker has decided to de-escalate medical care (patients with Do Not Resuscitate order but for whom standard care is continued will not be excluded)
* Known allergy to phenylephrine or norepinephrine
* Treated with vasopressor >12 hours for current episode of shock
* Preference of specific vasopressor agent by patient's provider
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj Keriwala, MD, MPH, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phenylephrine | Norepinephrine
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenylephrine | Norepinephrine | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Full Range); unit: years] | 63 [47 to 84] | 58.4 [47 to 73] | 60.4 [47 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17
Heart Rate [Mean (Full Range); unit: beats/minute] | 86.3 [60 to 119] | 97.3 [60 to 132] | 92.4 [60 to 132]
Mean Blood Pressure [Mean (Full Range); unit: mm/Hg] | 67.4 [51 to 95] | 66.2 [54 to 79] | 66.7 [51 to 95]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Heart Rate
Time Frame: Up to 28 days
Measure: Mean (Full Range); unit: beats/minute
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
beats/minute | 96.7 [65 to 132] | 108.6 [57 to 153]

2. Secondary Outcome: Number of Participants With Arrhythmia Events
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
Participants | 1 | 2

3. Secondary Outcome: Total Time in Arrhythmia
Time Frame: Up to 28 days
Population: only participants with arrhythmias included
Measure: Number; unit: minutes
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 1 | 2
minutes
  atrial fibrillation | 1224 | 209
  Other (undetermined) arrthymia | 0 | 2332

4. Secondary Outcome: Number of Patients With ST-segment Abnormalities on ECG
Description: ST Elevation of 1 mm in 2 or more consecutive leads or Horizontal or downsloping ST depression of 1 mm in 2 or more consecutive leads
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

5. Secondary Outcome: Number of Uses of Rate-controlling Agent
Description: includes use of Diltiazem, Esmolol, Metoprolol, Propranolol, Verapamil
Time Frame: Up to 28 days
Measure: Number; unit: number of uses
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
number of uses | 0 | 0

6. Secondary Outcome: Number of Times an Anti-arrhythmic Agent is Used
Time Frame: Up to 28 days
Measure: Number; unit: events
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
events | 2 | 1

7. Secondary Outcome: Use of Corticosteroid
Description: number of days participants received a corticosteroid
Time Frame: Up to 28 days
Measure: Number; unit: days
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
days | 1 | 10

8. Secondary Outcome: Number of Direct Current (DC) Cardioversion Events
Time Frame: Up to 28 days
Measure: Number; unit: DC cardioversion events
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
DC cardioversion events | 0 | 0

9. Secondary Outcome: Number of Days Mechanical Ventilation Needed
Time Frame: Up to 28 days
Population: only participants that required mechanical ventilation
Measure: Number; unit: days
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 2 | 6
days | 3 | 22

10. Secondary Outcome: Number of Days Hemodialysis Needed
Time Frame: Up to 28 days
Population: only participants that required dialysis
Measure: Number; unit: days
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 1 | 2
days | 1 | 11

11. Secondary Outcome: Mean Sequential Organ Failure Assessment (SOFA) Score
Description: Predicts ICU mortality based on lab results and clinical data. Range is 0-24 with higher numbers indicating a higher risk of mortality
Time Frame: Up to 28 days
Population: data was not collected
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants Developing Peripheral Limb Ischemia
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Cardiac Arrest Events
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

14. Secondary Outcome: Number of Days Without Vasopressor Use
Description: Shock free days
Time Frame: Up to 28 days
Measure: Number; unit: days
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
days | 154 | 151

15. Secondary Outcome: Number of Days Without Mechanical Ventilation
Description: Mechanical ventilation-free days
Time Frame: Up to 28 days
Measure: Number; unit: days
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
days | 165 | 164

16. Secondary Outcome: Days Without Dialysis
Description: Dialysis-free days
Time Frame: Up to 28 days
Measure: Number; unit: days
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
days | 168 | 152

17. Secondary Outcome: Hospital Days Not in ICU
Description: ICU free days
Time Frame: Up to 28 days
Measure: Number; unit: days
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
days | 144 | 139

18. Secondary Outcome: Days Spent Out of the Hospital
Description: Hospital free days
Time Frame: Up to 28 days
Measure: Number; unit: days
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
days | 103 | 98

19. Secondary Outcome: Readmission to ICU
Time Frame: Up to 28 days
Population: data was not collected
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Participants Rehospitalized After Discharge
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
Participants | 0 | 0

21. Secondary Outcome: Length of ICU Stay
Time Frame: Up to 28 days
Measure: Mean (Full Range); unit: days
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
days | 4.1 [2 to 6] | 5.2 [2 to 17]

22. Secondary Outcome: Length of Hospital Stay
Time Frame: Up to 28 days
Measure: Mean (Full Range); unit: days
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
days | 10 [4 to 26] | 8.9 [3 to 28]

23. Secondary Outcome: 28-day Mortality
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
Participants | 2 | 3

24. Secondary Outcome: Location of Death
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 1 | 4
Participants
  ICU | 0 | 4
  Not recorded | 1 | 0

25. Secondary Outcome: Cause of Death
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 2 | 3
Participants
  E. coli bacteremia, aspiration pnemonia | 0 | 1
  Respiratory failure,hospital aquired pneumonia | 1 | 0
  septic shock | 1 | 1
  Hypoxemic respiratory failure | 0 | 1

26. Secondary Outcome: Mean Troponin-I
Description: From chart review (if available)
Time Frame: Up to 28 days
Population: patients with troponin levels
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 1 | 2
ng/mL | 0.22 [0.22 to 0.22] | 0.38 [0.1 to 0.6]

27. Secondary Outcome: CK-MB
Description: From chart review (if available)
Time Frame: Up to 28 days
Population: patients with CK-MB levels
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 1 | 1
ng/mL | 8.87 [8.87 to 8.87] | 5.07 [5.07 to 5.07]

28. Secondary Outcome: Creatinine Kinase (CK)
Description: From chart review (if available)
Time Frame: Up to 28 days
Population: patients with CK levels
Measure: Mean (Full Range); unit: units/L
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 1 | 2
units/L | 738 [738 to 738] | 6986.6 [242 to 13211]

29. Secondary Outcome: Number of Participants Receiving Non-study Vasopressors
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
Participants | 3 | 3

30. Secondary Outcome: Amount of Time Non-study Vasopressors Used
Time Frame: Up to 28 days
Population: participants receiving non-study vasopressors
Measure: Number; unit: hours
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 3 | 3
hours
  Phenylephrine | 0 | 13
  Norepinephrine | 0 | 0
  Vasopressin | 8 | 22
  Epinephrine | 0 | 16

31. Other Pre Specified Outcome: Mean Blood Pressure (Maximum and Minimum)
Time Frame: Up to 28 days
Measure: Mean (Full Range); unit: mm/Hg
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
mm/Hg
  minimum | 55.8 [40 to 63] | 53.8 [42 to 65]
  maximum | 88.6 [77 to 109] | 79.5 [71 to 92]

32. Other Pre Specified Outcome: Mean Central Venous Pressure
Time Frame: Up to 28 days
Measure: Mean (Full Range); unit: mm/Hg
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 8 | 9
mm/Hg | 10.4 [7 to 14] | 11.7 [7 to 17]

33. Other Pre Specified Outcome: Mean Metabolic Panel Laboratory Values
Description: From chart review (if available)
Time Frame: Up to 28 days
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Mean Central Venous Oxygen Saturation
Description: From chart review (if available)
Time Frame: Up to 28 days
Population: patients with central venous pressure readings
Measure: Mean (Full Range); unit: mm/Hg
Arm/Group | Phenylephrine | Norepinephrine
Number analyzed (Participants) | 3 | 4
mm/Hg | 10.4 [7 to 14] | 11.7 [7 to 17]

35. Other Pre Specified Outcome: Anti-hypertensive Agents Used
Time Frame: Up to 28 days
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Diuretic Agents Used
Time Frame: Up to 28 days
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Inotropes Used
Time Frame: Up to 28 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse Events and Serious adverse events will not include organ failure or death that is related to septic shock, which are expected complications in this population, unless they are more severe than is expected or unusual in their happenstances.
Arm/Group | Phenylephrine | Norepinephrine
All-Cause Mortality (participants affected / at risk) | 2/8 | 3/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

LIMITATIONS AND CAVEATS:
Study was terminated early due to slow enrollment, lack of support and equipoise. PI left Vanderbilt and the record was completed with data recorded in REDCap.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes